CLINICAL TRIAL: NCT02577237
Title: Building Family Caregiver Skills Using a Simulation-based Intervention for Care of Patients With Head and Neck Cancer
Brief Title: Building Caregiver Skills Using a Simulation-based Intervention for Care of Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2315
Record Dates: First submitted 2015-10-14; First posted 2015-10-16 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Head and Neck Cancer
Keywords: caregiver; simulation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Caregiver education (Experimental): The intervention includes caregivers who will receive an education and support program throughout radiation treatment in addition to usual care by their doctors and nurses.
  Interventions: Behavioral: In-person education sessions; Other: Survey; Other: Interview
- Control Group: educational booklet (Active Comparator): The control group will receive an educational booklet about caregiving in addition to usual care by their doctors and nurses
  Interventions: Behavioral: NCI Booklet; Other: Survey; Other: Interview

INTERVENTIONS:
Behavioral: In-person education sessions — The intervention will be delivered by a radiation oncology nurse. Each of the four in-person sessions consists of approximately 30 minutes of educational content/simulation that addresses a specific caregiving topic and any issues or concerns that the caregiver may be experiencing.
  Other Names: intervention group; educational content/simulation
  Arms: Intervention Group: Caregiver education
Behavioral: NCI Booklet — Radiation Oncology Nurse will hand participant the NCI booklet
  Other Names: When Someone You Love is being Treated for Cancer
  Arms: Control Group: educational booklet
Other: Survey — written, qualitative assessments of areas including depression and anxiety, caregiver self-efficacy, care-giver self efficacy for head and neck cancer, health-related quality of life, patient performance status, demographics, and medical history.
Other: Interview — A structured series of open-ended questions will be used during a telephone interview with participants at four weeks post radiation treatment.
  Other Names: semi-structured interview; Open ended questions

SUMMARY:
Patients with head and neck cancer and their caregivers face many challenges. These include learning about cancer and its treatment, coping with symptoms from illness and treatment side effects, making adjustments to usual activities, and managing the emotional effects of having a serious illness. This study tests whether different forms of education and support can help family caregivers feel better prepared. To find out if education about caregiving and different kinds of support are effective, this study wants to compare approaches.One group includes caregivers who will receive an education and support program throughout radiation treatment in addition to usual care by their doctors and nurses. The other group receives an educational booklet about caregiving in addition to usual care by their doctors and nurses. The caregiver also completes surveys about his or her emotions, distress, confidence as a care giver, and quality of life. In addition, the study asks the caregiver questions about his or her age, race, ethnicity, marital status, employment status, education, annual household income, and current living arrangements. This pilot study will only be offered at the Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center Main Campus.

DETAILED DESCRIPTION:
Aim 1: Conduct a pilot test of the effects of a novel caregiver intervention, as compared to a control group, on family caregiver self-efficacy for caregiving, anxiety, depression, and health-related quality of life.

Aim 2: Explore the acceptability of a caregiver intervention that utilizes simulation.

Aim 3: Assess the feasibility of the intervention. Aim 4: Describe the incidence of patient events that may be impacted by caregiver self-efficacy, such as acute care visits, admissions to the hospital, visits to the emergency department, need for fluids in the radiation oncology department, and interrupted treatment course.

ELIGIBILITY:
Inclusion Criteria:

* family member or friend of an adult patient with a new diagnosis of Stage III - IV cancers of the tongue, gum, oral cavity, nasopharynx, oropharynx, hypopharynx, larynx, or parotid who is receiving radiation therapy for curative intent
* identified by the patient as his/her primary caregiver who is providing daily assistance and/or emotional support
* cognitively intact, as evidenced by orientation to person, place, and time
* ability to speak, read, and comprehend English

Exclusion Criteria:

* Caregivers of patients who are receiving hospice care will be excluded because of the patient's poor prognosis and multiple issues associated with end-of-life care
* Caregivers who are themselves undergoing active cancer treatment will be excluded (hormonal treatment allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Average efficacy of caregiving summary score | Up to 5 weeks
  Summary statistics as well as observed values of longitudinally measured efficacy outcome variables (efficacy for caregiving, anxiety, depression, and HRQOL) will be presented graphically. Linear mixed models will be used to estimate within- and between-subject components of variance needed for design of a larger trial with these endpoints.
Average anxiety summary score | Up to 5 weeks
  Summary statistics as well as observed values of longitudinally measured efficacy outcome variables (efficacy for caregiving, anxiety, depression, and HRQOL) will be presented graphically. Linear mixed models will be used to estimate within- and between-subject components of variance needed for design of a larger trial with these endpoints.
Average depression summary score | Up to 5 weeks
  Summary statistics as well as observed values of longitudinally measured efficacy outcome variables (efficacy for caregiving, anxiety, depression, and HRQOL) will be presented graphically. Linear mixed models will be used to estimate within- and between-subject components of variance needed for design of a larger trial with these endpoints.
Average Health Related Quality of Life (HRQOL) summary score | Up to 5 weeks
  Summary statistics as well as observed values of longitudinally measured efficacy outcome variables (efficacy for caregiving, anxiety, depression, and HRQOL) will be presented graphically. Linear mixed models will be used to estimate within- and between-subject components of variance needed for design of a larger trial with these endpoints.

SECONDARY OUTCOMES:
Qualitative assessment of acceptability | Up to 5 weeks
  Descriptive statistics will be used to summarize responses to semi-structured interviews
Attrition rate to assess feasibility | Up to 5 weeks
  Feasibility will be assessed via attrition and consent rates.
Consent rate to assess feasibility | Up to 5 weeks
  Feasibility will be assessed via attrition and consent rates.
Total time for delivering intervention to assess costs | Up to 5 weeks
  Time for delivering the intervention will be recorded to aid in assessing costs.
Average missed checklist items to assess integrity of intervention | Up to 5 weeks
  Integrity of the intervention will be assessed through monitoring of intervention checklist.
Event rate for patient events | Up to 5 weeks
  Describe the average incidence of all patient events that may be impacted by caregiver self-efficacy. Events may include acute care visits, admission to the hospital, visits to the emergency department, need for fluids in the radiation oncology department, and interrupted treatment course, and others

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mazanec, PhD, RN, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States